CLINICAL TRIAL: NCT01121120
Title: Phase II Study Evaluating the Safety and Efficacy of TXA127 in the Acceleration of Platelet Recovery Following Autologous Peripheral Blood Stem Cell Transplant in Patients With Hodgkin Lymphoma, Non-Hodgkin Lymphoma or Multiple Myeloma Undergoing Limited Reinfusion of CD34+ Cells
Brief Title: Acceleration of Platelet Recovery Following Autologous Peripheral Blood Stem Cell Transplant (PBSC) in Hodgkin, Non-Hodgkin Lymphoma or Multiple Myeloma Patients
Acronym: TXA127-PBSC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Tarix Pharmaceuticals (Industry)
Collaborators: Constant Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TXA127-2009-001
Record Dates: First submitted 2010-05-09; First posted 2010-05-12 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma
Keywords: Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple myeloma; Peripheral Blood Stem Cell Transplant; Autologous Peripheral Blood Stem Cell Transplant; Limited re-infusion of CD34+ cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TXA127 (Experimental): 300mcg/kg/day administered subcutaneously up to 28 days
  Interventions: Drug: TXA127
- Placebo (Placebo Comparator): 300mcg/kg/day administered subcutaneously up to 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TXA127 — 300mcg/kg/day, administered subcutaneously for up to 28 days
  Other Names: Angiotensin 1-7
  Arms: TXA127
Drug: Placebo — 300mcg/kg/day administered subcutaneously for up to 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of TXA127 in accelerating the time it takes for patients to recover their platelet counts following a Autologous Peripheral Blood Stem Cell transplant.

DETAILED DESCRIPTION:
* This is a randomized, double-blind (Investigator and Study Subject), placebo-controlled study.
* The conditioning regimen and mobilization agents used will be up to the discretion of the Study Center Investigator

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Subjects must have HL, NHL, or MM requiring PBSCT
* Subjects must have a life expectancy of at least 4 months
* Subjects are to receive autologous PBSC transplant following mobilization, CD34+ cells collected by apheresis, and conditioning chemotherapy
* Subjects must give written informed consent to participate in study. Consent must be obtained prior to the performance of any study-specific, non-institutional standard procedures. A copy of the signed informed consent will be retained in the subject's chart.
* Subjects must have CD34+ collection which allows reinfusion of ≥1.5 x 106 and ≤5.0 x 106 CD34+ cells/kg
* Subjects must have a psychological and emotional state that, in the view of the investigators, allows adherence to the protocol
* Female subjects capable of reproduction, and male subjects who have partners capable of reproduction, must agree to the following:

  * Use of an effective contraceptive method during the course of the study and for 2 months following the last administration of Investigational Product
  * Female subjects capable of reproduction must have a negative beta human chorionic gonadotropin (BHCG) serum or urine pregnancy test result within 7 days prior to first Investigational Product dose
  * Female subjects who are surgically sterilized or who have not experienced menses for at least two years are not required to have a pregnancy test

Exclusion Criteria:

* Subjects who have received radiotherapy to the pelvis and/or sternum within one year of first Investigational Product administration
* Subjects who have previously received or have planned Total Body Irradiation (TBI)
* Subjects with a history of prior malignancy other than HL, NHL, or MM that have not been in remission for >5 years, with the exception of basal cell or squamous cell carcinoma, cervical carcinoma in situ on biopsy, or localized prostate cancer (Gleason score <5)
* Subjects with a history of myelodysplastic syndrome
* Subjects who have had a venous or arterial embolic event AND who have received anti-coagulant treatment, where both the event and the treatment were within six months of the first Investigational Product administration
* Prior allogeneic hematopoietic cell transplant
* Presence of an uncontrolled infection or infection that required intravenous treatment within 7 days of entry
* Female subjects who are pregnant or breastfeeding
* Subjects who have received treatment with an investigational agent within 30 days of the projected first administration of Investigational Product (Day 0)
* Subjects with current alcohol use, illicit drug use, or any other condition (e.g., psychiatric disorder) that, in the opinion of the Investigator, may interfere with the subject's ability to comply with the study requirements or visit schedule
* Subjects with a known sensitivity to any of the Investigational Product components
* Subjects known to be seropositive for HIV or for HTLV-I
* Subjects for whom prophylactic platelet transfusions, at platelet counts >10× 109/L, are anticipated following PBSC transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Platelet recovery | ≤ 28 days from re-infusion of CD34+ cells
  Evaluate the effectiveness of TXA127 in accelerating the time to initial platelet recovery following PBSC transplant with a limited number of CD34+ cells, defined as CD34+ cell concentrations ≥1.5 x 106 and ≤5.0 x 106 CD34+ cells/kg. Platelet recovery is defined as that day the subject achieves a post-nadir platelet count of ≥20 x 109/L with no platelet transfusion in the prior 7 days.
Safety of TXA127 | ≤ 28 days from re-infusion of CD34+ cells
  Evaluate the safety of TXA127 administration following PBSC transplant

SECONDARY OUTCOMES:
Initial neutrophil recovery | ≤ 28 days from re-infusion of CD34+ cells
  Determine the effectiveness of TXA127 in accelerating the days to initial neutrophil recovery (ANCs > 0.5 x 10⁹/L)
Mucositis | ≤ 28 days from re-infusion of CD34+ cells
  Evaluate the incidence of mucositis Grade 3/4
Febrile neutropenia | ≤ 28 days from re-infusion of CD34+ cells
  Evaluate the effect of TXA127 in reducing the number of days of febrile neutropenia (fever and ANC <0.5 x 109/L)
Platelet transfusions | ≤ 28 days from re-infusion of CD34+ cells
  Evaluate the effect of TXA127 in reducing the number of platelet transfusions needed

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schuster, MD, Principal Investigator — Stony Brook university Medical Center
Locations (10):
- United States (10):
  - City of Hope Hospital, Duarte, California
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Stony Brook, Long Island City, New York
  - Montefiori Medical Center, The Bronx, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia